CLINICAL TRIAL: NCT06788431
Title: A Randomized, Double-blind, Placebo-controlled, Multiple-dose Escalation IIT Clinical Study to Evaluate the Efficacy and Safety of Injectable IMC-001 in Patients With Recent Acute Coronary Syndrome (ACS) Who Are Receiving Optimal Medical Therapy After PCI Treatment
Brief Title: A Study Evaluating the Stability and Efficacy of IMC-001 for Injection on Atherosclerotic Plaques in Patients With ACS.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Collaborators: RenJi Hospital (Other); ImmuneCare Biopharmaceuticals (Shanghai) Co., Ltd. (Other); The First Affiliated Hospital of Nanyang Medical College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMC-001-01
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Atherosclerosis
Keywords: Acute coronary syndrome; atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Acute Coronary Syndrome | interventions — IMC-001

STUDY DESIGN:
Intervention Model Description: Fifteen subjects were enrolled in each dose group, including 10 in the experimental group and 5 in the control group. The experimental group received IMC-001 and optimal drug treatment, and a total of 20 subjects were included, and the control group was given placebo and optimal drug treatment, and a total of 10 subjects were included
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMC-001 and Optimal medical treatment (Experimental)
  Interventions: Drug: IMC-001 and Optimal medical treatment
- IMC-001 placebo and Optimal medical treatment (Placebo Comparator)
  Interventions: Drug: IMC-001 placebo and optimal medical treatment

INTERVENTIONS:
Drug: IMC-001 and Optimal medical treatment — Subjects receive IMC-001 administered by injection and also receive optimal medical treatment.
  Arms: IMC-001 and Optimal medical treatment
Drug: IMC-001 placebo and optimal medical treatment — Subjects receive IMC-001 placebo administered by injection and also receive optimal medical treatment.
  Arms: IMC-001 placebo and Optimal medical treatment

SUMMARY:
A randomized, double-blind, placebo-controlled, multiple-dose escalation IIT clinical study to evaluate the efficacy and safety of injectable IMC-001 in patients with recent acute coronary syndrome (ACS) who are receiving optimal medical therapy after PCI treatment. Two dose groups, Fifteen subjects were enrolled in each dose group, including 10 in the experimental group and 5 in the control group. The experimental group received IMC-001 and optimal drug treatment, and a total of 20 subjects were included, and the control group was given placebo and optimal drug treatment, and a total of 10 subjects were included.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years old, male or female;
2. Patients with recent (within 30 days prior to enrollment) who have had acute coronary syndrome;
3. CTA examination of the presence of at least one measurable target vessel segment in the coronary artery, and the following two conditions must be met at the same time: the total volume of plaques with calcified volume accounting for <50%, and the presence of low-density attenuated plaques (LAP) that meet the definition of CTA;
4. High sensitivity C-reactive protein (hsCRP) ≥2.0 mg/L;
5. Subjects should take effective contraceptive measures to avoid pregnancy or impregnation of their partner during the period of taking the study drug until 6 months after stopping the drug;
6. Subjects understand and comply with the study process, participate voluntarily, and sign the informed consent form..

Exclusion Criteria:

Subjects who meet any of the following criteria cannot enter this study:

1. Those who have had cerebral infarction or TIA within the past 12 months.
2. Myocardial infarction within the previous 12 months (excluding acute myocardial infarction within 1 month before this dosing).
3. Previous treatment such as CABG, PCI, heart transplantation, SAVR/TAVR (patients who underwent PCI with ACS in the past three months can be included); or patients who are scheduled to undergo CABG, PCI, heart transplantation, SAVR/TAVR, etc. during the study period.
4. Recurrent arrhythmias with severe symptoms and ineffective drug treatment within the past 3 months, such as ventricular tachycardia, atrial fibrillation with rapid ventricular rate, and paroxysmal supraventricular tachycardia.
5. ECG showing QT prolongation, i.e., QTc interval ≥450ms in males and 470ms ≥ females, or family history of long QT syndrome (grandparents, parents, and siblings).
6. New York Heart Association (NYHA) Class III and above congestive heart failure.
7. History of arterial thrombosis or deep vein thrombosis within 6 months prior to enrollment, or history of spontaneous bleeding of any severity within 2 months prior to enrollment.
8. Active lung disease, including but not limited to interstitial lung disease or pneumonia, pulmonary fibrosis, etc.
9. Serious infection within 4 weeks prior to the first dose or active infection at screening, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonitis.
10. Abnormal laboratory indicators include, but are not limited to: neutrophils <1.5×109/L, hemoglobin <100 g/L, platelet count ≤100×109/L, total bilirubin >1.5× ULN, international normalized ratio (INR) >2× or activated partial thromboplastin time (APTT) >2× ULN, aspartate aminotransferase (AST) >2× ULN and alanine aminotransferase (ALT) >2× ULN , blood creatinine > 1.5× ULN.
11. Known previous allergy to macromolecular protein preparations/monoclonal antibodies, known allergy to the investigational drug or its excipients, or the same type of drug.
12. Those who have donated blood or lost ≥ 400 mL of blood within 3 months prior to dosing, received blood transfusion or used blood products.
13. Participated in any drug clinical trial or medical device clinical trial within 3 months before screening.
14. Those who have undergone major surgery within 3 months before screening or are expected to have major surgery during this study, including the screening period (except for patients who underwent PCI within the past 3 months).
15. Previous malignancy within the past 3 years, with the exception of basal or squamous cell skin cancer that has undergone curative treatment, superficial bladder cancer, carcinoma in situ of the cervix or breast, or other malignancies with low risk of metastasis and death (5-year survival >90%).
16. Vaccination with live or attenuated vaccines within 28 days before the first dose. But inactivated vaccines are available.
17. Hepatitis B surface antigen (HBsAg) positive, hepatitis B core antibody (HBcAb) positive, and HBV DNA titers outside the normal range (HBcAb-positive patients need regular HBV DNA testing and antiviral prophylaxis); Positive hepatitis C virus antibody and positive HCV-RNA; Human immunodeficiency virus (HIV) seropositive. Treponema pallidum antibody (TP-Ab) positive (if the Treponema pallidum serology test is positive, further non-Treponema pallidum serology test, which is negative and judged by the investigator to be cured of previous syphilis infection is eligible for inclusion).
18. Subjects with a history of drug abuse, alcohol abuse (alcohol abuse is defined as drinking 14 units of alcohol per week: 1 unit = 285mL of beer, or 25mL of spirits, or 100mL of wine).
19. Pregnant or lactating females; Positive pregnancy test during the screening period.
20. Subjects who are considered unsuitable for the study in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The change in low-attenuated plaque volume (LAPV) of the target vessel segment of the coronary artery was assessed by CT angiography (CTA). | Day 92 Day 176

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, M.D., Principal Investigator — RenJi Hospital
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Renji Hospital,Shanghai, Shanghai, Shanghai Municipality